CLINICAL TRIAL: NCT06659185
Title: Carbohydrate Mouth Rinsing and Softball Batting Performance: a Double-blind Crossover Study
Brief Title: Carbohydrate Mouth Rinsing and Softball Batting Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Chih-Hui Chiu, Professor, National Taiwan Sport University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 113-8
Record Dates: First submitted 2024-10-22; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Carbohydrate
Keywords: batting accuracy; performance
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: a double-blind crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate mouth rinsing (Experimental): Carbohydrate mouth rinsing for 20 seconds with 25 ml of 6.4% maltodextrin
  Interventions: Dietary Supplement: Exercise
- placebo (Placebo Comparator): Mouth rinsing for 20 seconds with 25 ml of water
  Interventions: Dietary Supplement: Exercise

INTERVENTIONS:
Dietary Supplement: Exercise — The effects of placobo mouth rinsing on softball batting performance
  Other Names: plocabo mouth rinsing

SUMMARY:
Participants rinsed their mouths for 20 seconds with 25 ml of either 6.4% maltodextrin (CMR) or placebo (PLA). After rinsing, the grip force, counter-movement jump (CMJ) and batting tests were performed in sequence.

DETAILED DESCRIPTION:
The purpose of this study was to investigate the effect of CMR on softball batting performance. Fourteen trained collegiate female softball players completed two trials in a randomization crossover trail, in which they rinsed their mouths for 20 seconds with 25 ml of either 6.4% maltodextrin (CMR) or placebo (PLA). After rinsing, the grip force, counter-movement jump (CMJ) and batting tests were performed in sequence. The tanner tee was utilised to perform five sets of five balls at a time, with a minimum of 3 minutes rest between sets. The batting test recorded average exit velocity, maximum exit velocity and batting accuracy. The standardized standard deviation (SD) for launch angle represents standardized variability.

ELIGIBILITY:
Inclusion Criteria:

* more than 6 years of professional fast-pitch softball training
* more than 6 months of continuous training
* from at least the top four teams in the country

Exclusion Criteria:

* non-professionally fast-pitch softball training
* lack of regular training in the past 6 months
* in the event that the applicant has sustained a sports injury or is currently experiencing epilepsy, hypertension, hyperlipidemia, heart disease, arthritis, osteoporosis, or a brain injury, and has yet to undergo a period of recuperation exceeding three months

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
exit velocity | 20 seconds after rinsing
  The average exit velocity

SECONDARY OUTCOMES:
batting accuracy | 20 seconds after rinsing
  The standardized standard deviation (SD) for launch angle represents standardized variability

CONTACTS AND LOCATIONS:
Overall Officials: Chih Hui Chiu, PhD, Principal Investigator — National Taiwan University of Sport
Locations (1):
- National Taiwan University of Sport, Taichung, North, Taiwan

IPD SHARING:
Plan to Share IPD: No
no share plan

DOCUMENTS (1):
  • Study Protocol (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT06659185/Prot_000.pdf